CLINICAL TRIAL: NCT05053659
Title: Phase I Trial of Loncastuximab Tesirine and Venetoclax for Treatment of Relapsed/ Refractory Non-Hodgkin Lymphoma
Brief Title: Loncastuximab Tesirine and Venetoclax for Relapsed/ Refractory Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Paolo Caimi, MD (Other)
Responsible Party: Sponsor-Investigator, Paolo Caimi, MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE5420
Record Dates: First submitted 2021-08-18; First posted 2021-09-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Relapsed Non Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — loncastuximab tesirine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Loncastuximab tesirine & venetoclax (Experimental): Participants will receive a baseline disease assessment via PET/CT in FDG avid lymphomas; CT scan (chest, abdomen, pelvis; inclusion of neck in selected cases). Bome marrow biopsy in selected cases.
  Premedication includes:
  * Allopurinol (to reduce uric acid) 300mg orally daily starting day -1 and continuing at least until day 7 of each cycle.
  * Dexamethasone (steroid pre-medication) 4mg orally twice daily on day -1, day 1 and day 2 of each cycle.
  * Adequate oral hydration starting on day -1 or -2, defined as 1 - 2 liters of oral intake of liquids in 24 hours
  Study treatment to be given every 21 days.
  * Loncastuximab tesirine (50 - 150 μg/kg) intravenously (IV) on day 1 of each 21-day cycle
  * Venetoclax (400 - 800 mg) orally, every day on days 1 - 5 of each 21-day cycle. Dose ramp-up on cycle 1 (over days 1 - 5 for target dose 400mg, 1 - 6 for target dose 600mg and 1 - 7 for target dose 800mg
  Interventions: Drug: Loncastuximab tesirine; Drug: Venetoclax

INTERVENTIONS:
Drug: Loncastuximab tesirine — Loncastuximab tesirine 50 - 150 μg/kg will be administered as a 30 minutes IV infusion on Day 1 of each cycle for 6 cycles. On doses over 100 μg/kg, subsequent dosing (i.e. beyond 100 μg/kg) will be done at 50% of the dose that is administered on the first 2 cycles.
  Other Names: ADCT-402; lonca
Drug: Venetoclax — Participants will receive venetoclax at target doses of 400 - 800mg orally on days 1 - 5 of each (21 day) cycle.
  On cycle 1, venetoclax dose will be escalated to reach the target dose over the course of 5 days for target dose 400mg, 6 days for target dose 600mg and 7 days for target dose 800mg
  Venetoclax should preferably be given after a meal and on cycle 1 should be preceded by prophylaxis for tumor lysis syndrome (TLS).
  Other Names: ABT-199; GDC-0199

SUMMARY:
The purpose of this study is to determine the correct dose and safety of combining two new cancer drugs, loncastuximab tesirine and venetoclax, as a treatment for relapsed or refractory B cell lymphoma.These drugs are used to treat some lymphomas, but have not yet been tested in combination for the treatment of lymphoma. The main goal of this study is to determine the safety of the combination.

DETAILED DESCRIPTION:
This is a phase I trial designed to evaluate the safety and tolerability of loncastuximab tesirine given in combination with venetoclax for treatment of relapsed/refractory non - Hodgkin lymphoma.

Loncastuximab tesirine is an investigational (experimental) drug that works by targeting a protein in cancer cells (called CD19) and delivering a small amount of chemotherapy directly to the cancer cells. Loncastuximab tesirine is experimental because it is not approved by the Food and Drug Administration (FDA). Venetoclax, is a targeted anti-cancer drug, which works by imitating a particular protein produced by the tumor and interrupting its normal processes, ultimately causing the tumor cells to die. Adding venetoclax to the loncastuximab tesirine regimen is believed to increase the chance of getting relapsed or refractory B cell lymphoma cancer in remission. Venetoclax is approved by the FDA for treatment in some types of cancer, but is not approved by the FDA for the treatment of lymphoma soit is considered experimental in this study. Up to 36 subjects will take in this phase I research study.

The primary objective for this study: To determine the safety and tolerability of the combination of loncastuximab tesirine and venetoclax to identify the recommended phase 2 dose (RP2D) of these agents.

Secondary objectives are:

* To describe the adverse event profile of the combination of loncastuximab tesirine and venetoclax.
* To describe the overall response rate (ORR) and complete response rate (CRR) of relapsed/refractory non-Hodgkin lymphoma treated with the combination of loncastuximab tesirine and venetoclax.
* To describe the overall survival (OS) and progression free survival (PFS) of subjects with relapsed / refractory non-Hodgkin lymphoma treated with the combination of loncastuximab tesirine and venetoclax.
* To describe the disease-free survival, the disease specific survival and time to treatment failure of subjects with relapsed/refractory non-Hodgkin lymphoma treated with the combination of loncastuximab tesirine and venetoclax.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologic or cytologic diagnosis of non-Hodgkin lymphoma, with the exclusion of small lymphocytic lymphoma/chronic lymphocytic leukemia.

  --Patients with mantle cell lymphoma are not eligible for the dose escalation part of the study. Inclusion of patients with mantle cell lymphoma to the dose expansion part of the study will be done after an amendment delineates a MCL - specific venetoclax ramp up and tumor lysis syndrome prophylaxis and monitoring regimen.
* Participants must have received ≥2 prior systemic therapies for their lymphoma.
* Participants must have measurable disease as defined by the 2014 Lugano Classification.
* Participants must meet clinical indications for treatment.
* ECOG performance status ≤ 2 (see Appendix I)
* Adequate bone marrow function, defined by the following laboratory parameters

  * Absolute neutrophil count of 1.0 x 109/L
  * Platelet count of 75 x 109/L; platelet count of 50 - 75 x 109/L are permitted in participants with marrow involvement by the lymphoma. Platelets must not have received a platelet transfusion in 7 days.
* Adequate organ function, defined by the following laboratory parameters

  * Adequate hepatic function, with transaminases (alanine aminotransferase [ALT], aspartate aminotransferase [AST], and gamma glutammyltransferase [GGT]) ≤ 2.5 times the upper limit of normal;
  * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
  * Calculated creatinine clearance > 30 mL/min by the Cockcroft-Gault equation.
  * For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 30 days after the last dose of venetoclax and at least 9 months after the last dose of loncastuximab tesirine for women.
  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (< 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).

Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

-For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

--With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose of loncastuximab. Men must refrain from donating sperm during this same period.

With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the last dose of loncastuximab to avoid exposing the embryo.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* Prior treatment toxicities not resolved to grade <2 according to NCI CTCAE 5.0 (with the exception of alopecia or grade 2 sensory peripheral neuropathy).
* Patients with spontaneous tumor lysis syndrome.
* Autologous stem cell transplant within 30 days of start of study drug (C1D1).
* Allogeneic stem cell transplant within 60 days of start of study drug (C1D1).
* Women who are pregnant or breastfeeding.
* Active graft versus host disease
* Active autoimmune disease
* Known seropositive and requiring anti-viral therapy for human immunodeficiency (HIV) virus. Note: Testing is not mandatory to be eligible.
* Malabsorption syndrome or other condition that precludes enteral route of administration.
* Known allergy to both xanthine oxidase inhibitors and rasburicase. Allergy to only one of these agents does not constitute an exclusion criterion.
* Use of strong CYP3A inhibitors or inducers.

  • All medications that fall in these categories should be discontinued 14 days or 5 half-lives, whichever is longer, prior to the first dose of study drug.
* Administration or consumption of any of the following within 3 days prior to the first dose of study drug:

  * Grapefruit or grapefruit products
  * Seville oranges (including marmalade containing Seville oranges)
  * Star fruit
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  * Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
  * Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative-, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate.
  * Other uncontrolled conditions including uncontrolled cardiovascular disease or arrythmia, decompensated diabetes or COPD.
  * Congenital long QT syndrome or a Fridericia correction of the QT measure (QTcF) interval of > 480 ms at screening (unless secondary to pacemaker or bundle branch block)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) during cycle 1 of loncastuximab tesirine and venetoclax | Up to Day 21
  Number of DLTs during cycle 1 (21 days) of loncastuximab tesirine and venetoclax
Maximum tolerated dose (MTD) of loncastuximab tesirine and venetoclax | 6 weeks
  Number of MTDs of loncastuximab tesirine and venetoclax

SECONDARY OUTCOMES:
Overall response rate (ORR) as measured by proportion of participants with Complete Response (CR) and Partial Response (PR) | Day 5 of cycle 1 (each cycle is 21 days)
  ORR, described as proportion of participants with CR and PR. Response assessed via Revised Response Criteria for Malignant Lymphoma
Overall response rate (ORR) as measured by proportion of participants with CR or PR | Between cycle 3 and 4 (21-day cycles) +/- 7 days
  ORR, described as proportion of participants with CR and PR. Response assessed via Revised Response Criteria for Malignant Lymphoma
Overall response rate (ORR) as measured by proportion of participants with CR or PR | End of treatment, aproximately day 84 +/- 7 days
  ORR, described as proportion of participants with CR and PR. Response assessed via Revised Response Criteria for Malignant Lymphoma
Overall response rate (ORR) | Followup, every 3 months up to one year after end of treatment
  ORR, described as a proportion. Response assessed via Revised Response Criteria for Malignant Lymphoma
Complete response rate (CRR) as measured by proportion of participants with CR | Day 5 of cycle 1 (each cycle is 21 days)
  ORR, described as a proportion. Response assessed via Revised Response Criteria for Malignant Lymphoma
Complete response rate (CRR) | Between cycle 3 and 4 (21-day cycles) +/- 7 days
  ORR, described as a proportion. Response assessed via Revised Response Criteria for Malignant Lymphoma
Complete response rate (CRR) | End of treatment, aproximately day 84 +/- 7 days
  ORR, described as a proportion. Response assessed via Revised Response Criteria for Malignant Lymphoma
Complete response rate (CRR) | Followup, every 3 months up to one year after end of treatment
  ORR, described as a proportion. Response assessed via Revised Response Criteria for Malignant Lymphoma
Overall survival (OS) | At end of follow-up (1 year)
  OS is defined as the time from the date of study entry to the date of death, with censoring done on live patients at the time of last follow up. OS will be estimated using the Kaplan Meier method
Progression free survival (PFS) | At end of follow-up (1 year)
  PFS is defined as the time from entry onto study until lymphoma progression or death from any cause. PFS will be estimated using the Kaplan Meier method
  The precise date of progression is generally unknown. It may be defined as the first date of documentation of a new lesion or enlargement of a previous lesion, or the date of the scheduled clinic visit immediately after radiologic assessment has been completed. Where there is missing information, censoring of the data may be defined as the last date at which progression status was adequately assessed or the first date of unscheduled new anti-lymphoma treatment.
Median disease-free survival | At end of follow-up (1 year)
  Disease-free survival is measured from the time of occurrence of disease-free state (e.g. the adjuvant setting following surgery or radiation therapy) or attainment of a complete remission) to disease recurrence or death from lymphoma or acute toxicity of treatment.
Median disease-specific survival | At end of follow-up (1 year)
  Disease-specific survival is defined as death from lymphoma, or from toxicity from the drug. Death from unknown causes should be attributed to the drug
Time-to-treatment failure | At end of follow-up (1 year)
  Time to treatment failure (event-free survival) is measured from the time from study entry to any treatment failure including discontinuation of treatment for any reason, such as disease progression, toxicity, patient preference, initiation of new treatment without documented progression, or death.
Total number of adverse events during and after treatment | At end of treatment (21-day cycles until disease progression or toxicity, up to 6 cycles max)
  The objective is to describe the adverse event profile of the combination therapy by reporting number of adverse events during and after treatment, described as a proportion
Duration of response (DOR) | At end of follow-up (1 year)
  DOR, as measured by the median time in months of from first response (PR or CR) until relapse or death, using Kaplan Meier
Time to Progression (TTP) | At end of follow-up (1 year)
  TTP as measured by median time in months from treatment to death or relapse
Partial response rate (PRR) | At end of follow-up (1 year)
  PRR, as measured by proportion of patients with partial response

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Caimi, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share Individual Participant Data (IPD)